CLINICAL TRIAL: NCT00005565
Title: Mechanisms of Low Levels of Apolipoprotein B
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5114; R01HL056895 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypobetalipoproteinemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypobetalipoproteinemias

SUMMARY:
To determine mechanisms of low levels of apolipoprotein B.

DETAILED DESCRIPTION:
BACKGROUND:

Elevated apoB levels are associated with an increased risk of coronary heart disease. Hypobetalipoproteinemia (HBLP) is characterized by apoB levels less than the 5 percentile. Dr. Welty, the principal investigator, sequenced mutations for truncated forms of apoB-67, apoB-55 and apoB-44.4 which causes HBLP, described a kindred from the Framingham Heart Study with HBLP due to an unidentified apoB gene mutation and purified apoB-67 containing lipoprotein particles. Heterozygous apoB-67 subjects have one normal allele making apoB-100; therefore, apoB levels would be predicted to be at least 50 percent of normal; however, they are 24 percent of normal. Dr. Welty has shown that these lower than expected levels result from decreased production of VLDL apoB-100, LDL apoB-100 and apoB-67, increased catabolism of VLDL apoB-100, and increased direct removal of apoB-67 from VLDL.

DESIGN NARRATIVE:

The first aim is to locate the apoB gene mutation in the Framingham kindred. The second aim is to perform stable isotope studies in the apoB-55 and apoB-44.4 kindreds to determine if apoB metabolism for these shorter truncations is similar to that for apoB-67. In aim three, apoB-100 synthesis is studied in heterozygous apoB-70 transgenic mice. If it is 25-25 percent of normal litter mates, the mechanism for this reduction in apoB-100 levels will be studied in hepatocytes isolated from the transgenic mice. In specific aim 4, size and composition of VLDL are compared in apoB-67 subjects and controls to determine if larger size or compositional changes account for the faster catabolism of VLDL apoB-100. The study has been extended through June 2007.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-08; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Welty — Beth Israel Deaconess Medical Center

REFERENCES:
- [Background] Welty FK, Lichtenstein AH, Barrett PH, Dolnikowski GG, Schaefer EJ. Human apolipoprotein (Apo) B-48 and ApoB-100 kinetics with stable isotopes. Arterioscler Thromb Vasc Biol. 1999 Dec;19(12):2966-74. doi: 10.1161/01.atv.19.12.2966. PMID 10591677
- [Background] Welty FK, Lichtenstein AH, Barrett PH, Jenner JL, Dolnikowski GG, Schaefer EJ. Effects of ApoE genotype on ApoB-48 and ApoB-100 kinetics with stable isotopes in humans. Arterioscler Thromb Vasc Biol. 2000 Jul;20(7):1807-10. doi: 10.1161/01.atv.20.7.1807. PMID 10894821
- [Background] Welty FK, Guida KA, Andersen JJ. Donor splice-site mutation (210+1G_C) in the ApoB gene causes a very low level of ApoB-100 and LDL cholesterol. Arterioscler Thromb Vasc Biol. 2001 Nov;21(11):1864-5. No abstract available. PMID 11701479
- [Background] Matthan NR, Welty FK, Barrett PH, Harausz C, Dolnikowski GG, Parks JS, Eckel RH, Schaefer EJ, Lichtenstein AH. Dietary hydrogenated fat increases high-density lipoprotein apoA-I catabolism and decreases low-density lipoprotein apoB-100 catabolism in hypercholesterolemic women. Arterioscler Thromb Vasc Biol. 2004 Jun;24(6):1092-7. doi: 10.1161/01.ATV.0000128410.23161.be. Epub 2004 Apr 15. PMID 15087307
- [Background] Welty FK, Lichtenstein AH, Barrett PH, Dolnikowski GG, Schaefer EJ. Interrelationships between human apolipoprotein A-I and apolipoproteins B-48 and B-100 kinetics using stable isotopes. Arterioscler Thromb Vasc Biol. 2004 Sep;24(9):1703-7. doi: 10.1161/01.ATV.0000137975.14996.df. Epub 2004 Jul 8. PMID 15242863